CLINICAL TRIAL: NCT01723657
Title: Risk Adapted Treatment for Primary AML in Adults, Based on Genetics and Minimal Residual Disease (MRD) in Patients up to the Age of 70 Years.
Brief Title: Risk Adapted Treatment for Primary Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-03
Record Dates: First submitted 2012-10-31; First posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Leukemia; Myeloid; Acute; Young; CETLAM
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risk-adapted postremission treatment. (Other): Ara-C, G-CSF, Autologous peripheral blood stem cell transplantation, Allogeneic matched related or unrelated donor transplant, G-CSF Priming, CD34+ selection, Myeloablative or reduced intensity conditioning, Mylotarg purging before autologous PBSC transplantation.
  Interventions: Drug: Ara-C; Other: Autologous peripheral blood stem cell transplantation.; Other: Allogeneic matched related or unrelated donor transplant.; Drug: G-CSF; Other: CD34+ selection.; Other: Mylotarg purging before autologous PBSC transplantation

INTERVENTIONS:
Drug: Ara-C — * Intermediate dose during induction phase to remission.
  * High dose during consolidation phase in patients with favorable cytogenetics and leukocyte index below 20.
Other: Autologous peripheral blood stem cell transplantation. — * In patients with favorable cytogenetics with a Leukocyte index above 20.
  * Patients with normal karyotype, and one cycle of chemotherapy to achieve complete remission, without adverse molecular and/or minimal residual disease (MRD) characteristics, regardless availability of a matched donor.
Other: Allogeneic matched related or unrelated donor transplant. — -Patients without favorable/intermediate characteristics.
Drug: G-CSF — * Administration at induction phase to remission, days 0 to 7. G-CSF will not be initiated if the leukocyte count is over 30x10e9/L at diagnosis or will be interrupted if the leukocyte count during treatmen arises 30x10e9/L.
  * Administration at consolidation phase, days 4 to 6 (3 doses). G-CSF will be interrupted if the leukocyte count during treatment arises 30x10e9/L.
  Other Names: Filgastrim.
Other: CD34+ selection. — -Patients with adverse prognosis with allogeneic peripheral blood stem cell (PBSC)tranplantation, CD34+ cell selection of the inoculum was performed.
Other: Mylotarg purging before autologous PBSC transplantation — Patients without favorable/intermediate characteristics and without matched related donor.

SUMMARY:
The AML-03 regimen investigates the addition of G-CSF priming to both induction and consolidation chemotherapies administrated in the previous AML-99 trial (NCT01716793) refines risk-stratification based on biological characterization also the AML-03 trial incorporates novel approaches for hematopoietic stem cell transplantation: such as Mylotarg™ "in vivo purging" in autografts, extends unrelated volunteers donors for allotransplants in high-risk patients, and introduces reduced intensity conditioning in patients with elder age (more than 50 years old).

The aims of these modifications are to analyse eficacy and toxicity of this induction and consolidation therapy and to analyse the disease free survival in patients who achieved complete response following a risk adjusted therapy.

DETAILED DESCRIPTION:
Induction chemotherapy: idarubicin (12mg/m2/day intravenous, days 1, 3 and 5), intermediate-dose cytarabine (500mg/m2/12h, intravenous, days 1, 3 and 5) and etoposide (100mg/m2/day, intravenous, from day 1 to 3) as in AML-99 trial (NCT01716793), with the addition of subcutaneous G-CSF from day 0 to the last day of chemotherapy. This induction therapy is repeated if complete remission (CR) is not achieved after the first course of treatment.

Consolidation therapy (as in AML-99 trial): mitoxantrone (12mg/m2/day, intravenous, days 4 to 6) and intermediate-dose cytarabine (500mg/m2/12h from day 1 to 6).

Risk-stratification according to cytogenetics, courses to CR and availability of an HLA-identical sibling:

* Patients in the favorable cytogenetics group [t(8;21), inv(16) or t(16;16)] and Leukocyte index <20 at diagnosis (LI=white blood cell count (WBC) x (blasts in bone marrow/100) are treated with one course of high-dose cytarabine (3g/m2/12h, intravenous, days 1, 3 and 5), but in case of LI>20 at diagnosis the intention is to perform an autologous peripheral blood stem cell (PBSC) transplantation.
* Patients in intermediate risk group, with normal karyotype, a single course of induction chemotherapy to achieve the CR, the absence of adverse molecular features (FLT3-ITD or MLL-PTD) and low minimal residual disease levels after consolidation (MRD<0,1%) receive an autologous PBSC transplant, regardless of having an HLA-identical sibling.
* The remaining patients defined as high-risk patients are treated with an allogeneic stem cell transplantation. Depending on the age, if the patient has an HLA-identical sibling donor, up to age of 50 years old it is performed with conventional conditioning therapy and positive selection of CD34+, older patients receive a reduced intensity conditioning regimen.
* Very high risk patients without a sibling are allocated to unrelated donor (9-10/10). Patients with adverse cytogenetics and/or FLT3-ITD without an adequate donor received Mylotarg™ as "in vivo purging" followed by an autologous PBSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML, classified using OMS criteria.
* Patients with 70 years old or younger.

Exclusion Criteria:

* Patients previously treated for the AML with chemotherapy different from hidroxiurea.
* Acute promyelocytic leukemia with t(15;17).
* Cronic mieloid leukemia in blastic crisis.
* Leukemias that appear after other myeloproliferative processes.
* Leukemias that survive after myelodysplasic syndromes of more than 6 months of evolution.
* Presence of other neoplasic disease in activity.
* Secondary AML which appears after cured malignant disease (for instance, Hodgking disease), and those who are still exposed to alkilant agents or radiation.
* Abnormal renal and hepatic functions with creatinin and/or bilirrubine 2 times higher than the normal threshold, except when the alteration should be attributed to the leukemia.
* Patient with an ejection fraction below 40%, symptomatic cardiac deficiency or both.
* Patients with neurological or concomitant psychiatric disease.
* Positivity by HIV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2003-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Complete remission rate (CRR) | 2 months.
  Analyze the efficacy and toxicity of IDICE-G (idarubicin, intermediate doses of ara-C and etoposide) and G-CSF to achieve complete remission.
Disease free survival (DFS). | 4 years.
  Analyze the disease free suvival of patients in remission, with a therapeutic strategy adjusted to the prognostic factors.
  Mortality in remission after chemotherapy and/or peripheral blood stem cell tranplantation.

SECONDARY OUTCOMES:
Toxicity in patients over 60 years old. | 4 years.
  Toxicity of the induction and intensification treatment in patients with more than 60 years old, in terms of unexpected adverse drug reaction, morbidity and mortality.
Evaluation of minimal residual disease (MRD) by flow cytometry and/or molecular markers during and after treatment. | 4 years.
  Study the immunophenotype characteristics and/or molecular markers at diagnosis, and during the different treatment phases.
Feasibility of post-remission treatment in patients with 60 or more years old. | 4 years.
  Study the effect of post-remission treatments in patients with more than 60 years to evaluate the success of consolidation treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sierra, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Salut Brunet, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (21):
- Spain (21):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Centro Medico Teknon, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - ICO Hospital Universitari de Bellvitge, L'Hospitalet Del Llobregat, Barcelona
  - Hospital A Coruña, A Coruña, Coruña
  - Hopital Universitari de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitari Son Dureta, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Murcia, Murcia, Murcia
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Universitari Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Mutua de Terrassa, Terrassa, Terrassa
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid, Valladolid